CLINICAL TRIAL: NCT02730767
Title: Effects of a 1-year Partially Supervised Exercise Program in Childhood Cancer Survivors - a Randomized Controlled Trial
Brief Title: SURfit - A Physical Activity Intervention for Childhood Cancer Survivors
Acronym: SURfit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SURfit
Record Dates: First submitted 2015-12-10; First posted 2016-04-06 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Late-effects of Childhood Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Partially supervised exercise intervention: Survivors in the intervention group will be asked to add at least 2.5 hours of intense physical activities per week. These should include at least 30 min of strength building exercises and 2 hours of aerobic exercises per week. Exercise bouts lasting 20 min or longer will be counted with respect to total weekly training time.
  Interventions: Behavioral: partially supervised exercise intervention
- Control Group (No Intervention): The control group will keep their physical activity level constant over the 1 year of the study. Thereafter, they will have the opportunity to receive the same intervention than the intervention group had received (off-trial) to benefit in the same way from an active lifestyle.

INTERVENTIONS:
Behavioral: partially supervised exercise intervention
  Other Names: physical activity intervention
  Arms: Intervention Group

SUMMARY:
Exercise can play a major role to mitigate or even prevent late effects in cancer survivors, such as cardiovascular disease, obesity, osteoporosis, fatigue, depression, reduced quality of life, mental health and physical performance.

The objective of this study is to assess the effect of an exercise program of 1 year on cardiovascular health, obesity and diabetes, osteoporosis, physical fitness, mental health and quality of life in childhood cancer survivors. The investigators will recruit childhood cancer survivors aged 16 years and above from three Swiss paediatric oncology clinics and randomize them into an intervention and a control group. The intervention group will be asked to increase physical activity for 1 year by at least 2.5 hours of intense physical activity weekly. Regular feedback will be given via a step counter, an online activity diary, and by the centre staff. The control group participants will keep their activity level constant. All participants will be seen after 3, 6 and 12 months to assess health and quality of life parameters over one year. After 1 year, the control group is offered to receive the same intervention to profit as well from an active lifestyle.

If the program shows to be effective, a complete package will become available to interested centres treating paediatric cancer patients in Switzerland to promote exercise in all survivors. The program will allow clinicians without previous experience in exercise counselling to improve the care of their patients.

ELIGIBILITY:
Inclusion Criteria:

* Registered in the Swiss Childhood Cancer Registry.
* Age at cancer diagnosis <16 years.
* Diagnosed with a cancer classifiable within the International Classification of Childhood Cancer (ICCC-3) or diagnosed with a Langerhans Cell Histiocytosis.
* Diagnosed and/or treated at the University Children's Hospital Basel, Cantonal Hospital of Aarau and/or Cantonal Hospital of Lucerne.
* Survived ≥5 years since primary cancer diagnosis or any subsequent cancer event (relapse or further cancer diagnoses)
* Age at the time of the study ≥16 years
* Informed Consent as documented by signature

Exclusion Criteria:

* Participation in another clinical trial <4 weeks prior to baseline assessment (eventually later re-enrolment)
* Contradiction to one of the inclusion criteria mentioned above
* Inability to exercise
* Exercise potentially harmful
* Women who are pregnant or breast feeding
* Women who intend to become pregnant during the course of the study
* Instable clinical condition (eventually later re-enrolment)
* Under treatment for relapse or further cancer diagnoses
* Cardiac arrhythmias under exercise (during baseline assessment or by history)
* Diagnosis of diabetes <3 months ago (eventually re-enrolment after 3 months if diabetes is under good control)
* Detection of a clinical condition that needs immediate treatment during baseline assessments (eventually re-enrolment after 3 months if in stable clinical condition)
* Planned relevant surgeries for the next 12 months
* Major musculoskeletal injuries, fractures <2 months ago (eventually later re-enrolment)
* Recent change in medication that interfere with the parameters of the CVD risk score (primary outcome) <1 month ago (eventually later re-enrolment)
* >4 hours of reported vigorous activities per week
* Inability to follow the procedures and understand the intervention and assessments of the study e.g. due to cognitive impairment, language problems, psychological disorders etc.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Composite cardiovascular risk score [z-score] | 12 months
  summarized mean z-score of waist circumference, blood pressure, HOMA-IR, inverted high density lipoprotein cholesterol, triglycerides and cardiorespiratory fitness

SECONDARY OUTCOMES:
Waist circumference [cm] | 3, 6, and 12 months
Systolic and diastolic blood pressure [mmHg] | 3, 6, and 12 months
Homeostasis Model Assessment Insulin Resistance (HOMA-IR) | 6 and 12 months
  calculated from insulin and glucose
HbA1C [mmol/mol] | 6 and 12 months
Insulin resistance from response to oral glucose tolerance test (oGTT) | 12 months
  Assessment of fasting glucose [mmol/l] and insulin [mIU/l] and glucose 2 hours after drinking of a glucose solution
Inverted high-density lipoprotein cholesterol (HDL) [mmol/l] | 6 and 12 months
Low-density lipoprotein cholesterol (LDL) [mmol/l] | 6 and 12 months
Total cholesterol [mmol/l] | 6 and 12 months
Triglycerides [mmol/l] | 6 and 12 months
Body Mass Index (BMI) [z-score] | 3, 6, and 12 months
  Calculated from height and weight
Absolute [kg] and relative [%] body fat mass | 3, 6, and 12 months
  Assessed with two methods: skinfold measurement (3, 6, and 12 months) and dual x-ray absorptiometry (DXA, 12 months only).
Areal bone mineral density [g/cm2 and z-scores] | 12 months
  Bone mineral density for total body, lumbar spine, and femoral neck assessed with dual x-ray absorptiometry (DXA)
Bone mineral content [g/cm and z-scores] | 12 months
  Bone mineral content for total body, lumbar spine, and femoral neck assessed with dual x-ray absorptiometry (DXA)
Total cross sectional bone area [mm2 and z-scores] | 12 months
  Cross sectional area of the distal and proximal sites of radius and tibia assessed with peripheral quantitative computer tomography (pQCT)
Cortical cross sectional bone area [mm2 and z-scores] | 12 months
  Cross sectional area of the proximal site of radius and tibia assessed with peripheral quantitative computer tomography (pQCT)
Total and trabecular bone mineral density [g/cm3 and z-scores] | 12 months
  Bone mineral density of the distal site of radius and tibia assessed with peripheral quantitative computer tomography (pQCT)
Cortical bone mineral density [g/cm3 and z-scores] | 12 months
  Bone mineral density of the proximal site of radius and tibia assessed with peripheral quantitative computer tomography (pQCT)
Muscle cross-sectional area [cm2 and z-scores] | 12 months
  Muscle cross-sectional area of the proximal site of radius and tibia assessed with peripheral quantitative computer tomography (pQCT)
Peak oxygen uptake (VO2max) [ml/(kg*min) and % predicted] | 6 and 12 months
  Assessed with maximal spiroergometry test
Peak performance [watt/kg and % predicted] | 6 and 12 months
  Assessed with maximal spiroergometry test
Heart rate recovery [delta beats/min] | 6 and 12 months
  Assessed at the end of the maximal spiroergometry test: delta beats/min between peak heart rate and heart rate 1 minute post exercise.
Hand grip strength in the left and right hand [kg] | 6 and 12 months
  Assessed with a hydrolic hand grip dynamometer.
Leg strength and endurance [repetitions/min] | 6 and 12 months
  Assessed with the 1 minute sit-to-stand test
Total physical activity [counts/min] | 6 and 12 months
  Assessed by accelerometer
Moderate to vigorous physical activities [minutes/day] | 6 and 12 months
  Assessed by accelerometer
High impact activities with ground forces >3.9 G [n/day] | 6 and 12 month
  Assessed by accelerometer
Sedentary behaviour [minutes/day] | 6 and 12 months
  Assessed by accelerometer
Number of steps per day [steps/day] | 6 and 12 months
  Assessed by accelerometer
Health related quality of life [T-score with mean=50, standard deviation=10 and range=0-100] | 6 and 12 months
  Health related quality of life assessed by the self-reported questionnaire short form 36 (SF-36).
Psychological distress [T-score with mean=50, standard deviation=10 and range=0-100] | 6 and 12 months
  Psychological distress assessed by the self-reported questionnaire Brief Symptom Inventory (BSI).
Fatigue on a visual analogue scale (VAS) [mm] | 3, 6 and 12 months
Fatigue | 3, 6 and 12 months
  Fatigue assessed with the self-reported questionnaire Checklist of Individual Strength (CIS).
Number of adverse events and serious adverse events [n] | 3, 6 and 12 months
  Number of participants with adverse events and exercise related complications categorized into seriousness of the event (adverse event [AE] or severe adverse event [SAE]).
Proportion of aimed physical activity reached [%] | 12 months
  Only intervention participants: compliance with intervention
Number of weeks where physical activity aim was reached [n/year] | 12 months
  Only intervention participants: compliance with intervention
Number of missing days in the online diary [n/year] | 12 months
  Only intervention participants: compliance with intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas X von der Weid, Prof, MD, Principal Investigator — University Children's Hospital Basel, UKBB
Locations (1):
- University Children's Hospital Basel (UKBB), Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rueegg CS, Zurcher SJ, Schindera C, Jung R, Deng WH, Banteli I, Schaeff J, Hebestreit H, von der Weid NX, Kriemler S. Effect of a 1-year physical activity intervention on cardiovascular health in long-term childhood cancer survivors-a randomised controlled trial (SURfit). Br J Cancer. 2023 Oct;129(8):1284-1297. doi: 10.1038/s41416-023-02410-y. Epub 2023 Aug 31. PMID 37653075
- [Background] Deng WH, Zurcher SJ, Schindera C, Jung R, Hebestreit H, Banteli I, Bologna K, von der Weid NX, Kriemler S, Rueegg CS. Effect of a 1-year physical activity intervention on quality of life, fatigue, and distress in adult childhood cancer survivors-A randomized controlled trial (SURfit). Cancer. 2024 May 15;130(10):1869-1883. doi: 10.1002/cncr.35207. Epub 2024 Feb 5. PMID 38315522
- [Background] Schindera C, Zurcher SJ, Jung R, Boehringer S, Balder JW, Rueegg CS, Kriemler S, von der Weid NX. Physical fitness and modifiable cardiovascular disease risk factors in survivors of childhood cancer: A report from the SURfit study. Cancer. 2021 May 15;127(10):1690-1698. doi: 10.1002/cncr.33351. Epub 2021 Jan 6. PMID 33405260
- [Background] Jung R, Zurcher SJ, Schindera C, Braun J, Deng WH, von der Weid NX, Rueegg CS, Kriemler S. Adherence and contamination in a 1-year physical activity program in childhood cancer survivors: A report from the SURfit study. Cancer Med. 2023 Jul;12(13):14731-14741. doi: 10.1002/cam4.6096. Epub 2023 May 18. PMID 37199378
- [Background] Jung R, Zurcher SJ, Schindera C, Eser P, Meier C, Schai A, Braun J, Deng WH, Hebestreit H, Neuhaus C, Schaeff J, Rueegg CS, von der Weid NX, Kriemler S. Effect of a physical activity intervention on lower body bone health in childhood cancer survivors: A randomized controlled trial (SURfit). Int J Cancer. 2023 Jan 15;152(2):162-171. doi: 10.1002/ijc.34234. Epub 2022 Aug 26. PMID 35913755
- [Background] Zurcher SJ, Jung R, Monnerat S, Schindera C, Eser P, Meier C, Rueegg CS, von der Weid NX, Kriemler S. High impact physical activity and bone health of lower extremities in childhood cancer survivors: A cross-sectional study of SURfit. Int J Cancer. 2020 Oct 1;147(7):1845-1854. doi: 10.1002/ijc.32963. Epub 2020 Mar 25. PMID 32167159
- [Background] Rueegg CS, Kriemler S, Zuercher SJ, Schindera C, Renner A, Hebestreit H, Meier C, Eser P, von der Weid NX. A partially supervised physical activity program for adult and adolescent survivors of childhood cancer (SURfit): study design of a randomized controlled trial [NCT02730767]. BMC Cancer. 2017 Dec 5;17(1):822. doi: 10.1186/s12885-017-3801-8. PMID 29207962
- [Derived] Schindera C, Usemann J, Zuercher SJ, Jung R, Kasteler R, Frauchiger B, Naumann G, Rueegg CS, Latzin P, Kuehni CE, von der Weid NX. Pulmonary Dysfunction after Treatment for Childhood Cancer. Comparing Multiple-Breath Washout with Spirometry. Ann Am Thorac Soc. 2021 Feb;18(2):281-289. doi: 10.1513/AnnalsATS.202003-211OC. PMID 32877212